CLINICAL TRIAL: NCT04821583
Title: Hydrocortisone Treatment for Symmetric Lipomatosis Associated With Neuropathy (SLN): an N-of-1 Study
Brief Title: Hydrocortisone Treatment for Symmetric Lipomatosis Associated With Neuropathy (SLN): an N-of-1 Study Hydrocortisone Treatment for Symmetric Lipomatosis Associated With Neuropathy (SLN): an N-of-1 Study
Acronym: N-of-1 SLN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, dr. Laura C. G. de Graaff-Herder, Principal investigator, Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-of-1 SLN
Record Dates: First submitted 2021-03-16; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Symmetric Lipomatoses, Multiple
Keywords: Symmetric Lipomatosis associated with Neuropathy; Hydrocortisone; Lipoma; Neuropathy
MeSH Terms: conditions — Lipomatosis, Multiple Symmetrical; Lipoma | interventions — Hydrocortisone

STUDY DESIGN:
Intervention Model Description: An N-of-1 study is considered as a reliable and suitable design to assess the efficacy of a treatment at an individual level. The study will consist of two cycles with each two periods of active treatment or placebo, a run-in period, tapering period and a wash-out period. Within each cycle, the sequence of the hydrocortisone and placebo period is randomized.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both the participant and the investigator are masked. The investigator is also the care provider and outcomes assessor. The statistician and clinical pharmacist are unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrocortisone (Experimental): Hydrocortisone (20 mg/day) in a 10-5-5 schedule: 10 mg at 0700h, 5 mg at 1200h, and 5 mg at 1700h. The hydrocortisone periods last 10 weeks per period. In total, there are two hydrocortisone periods.
  Interventions: Drug: Hydrocortisone
- Placebo (Placebo Comparator): Placebo (20 mg/day) in a 10-5-5 schedule: 10 mg at 0700h, 5 mg at 1200h, and 5 mg at 1700h. The placebo periods last 10 weeks per period. In total, there are two placebo periods.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrocortisone — Hydrocortisone is orally administered.
  Arms: Hydrocortisone
Drug: Placebo — Placebo is orally administered.
  Arms: Placebo

SUMMARY:
A young women with Symmetric Lipomatosis associated with Neuropathy (SLN) was seen at the department of Internal Medicine - Endocrinology and at the department of Neurology at the Erasmus MC, Rotterdam, the Netherlands. The patient presented with balance problems due to neuropathy and prominent cervical and genital lipomas. In the past, the patient had been treated with steroids for a short period. The patient noticed that, as a 'side effect', during this treatment period the lipomas shrank and that the balance problems nearly disappeared. The complaints reappeared after withdrawal of the steroids. In the current study, the usefulness of steroid treatment in this single patient will be investigated in an N-of-1 trial.

Primary objective: to determine the efficacy of hydrocortisone treatment for neuropathy on an individual level in a patient with SLN as assessed with the Rasch-built Overall Disability Scale (RODS).

DETAILED DESCRIPTION:
A young women with Symmetric Lipomatosis associated with Neuropathy (SLN) was seen at the department of Internal Medicine-Endocrinology and the department of Neurology at the Erasmus MC, Rotterdam, the Netherlands. SLN is a rare disorder characterized by symmetric lipomas and neuropathy due to a homozygous mutation of c.2119C>T p.R707W in the MFN2 gene. Only seven cases of SLN are known in the literature. The patient presented with balance problems due to neuropathy and prominent cervical and genital lipomas. In the past, the patient had been treated with steroids (prednisolone) for a short period, because of a suspicion of adrenal insufficiency. The patient noticed that, as a 'side effect', during this treatment period the lipomas shrank and that the balance problems nearly disappeared. However, as a synacthen test showed that adrenal function was normal, steroid treatment was tapered and the complaints reappeared. In a follow-up visit at our outpatient clinic, the patient requested to be treated again with steroids for the complaints. As there is no literature on the effects of treatment with steroids on balance problems and on the size of lipomas in patients with SLN, the usefulness of steroid treatment in this single patient is investigated in an N-of-1 trial in order to improve the clinical care for this patient.

Primary objective: to determine the efficacy of hydrocortisone treatment for neuropathy on an individual level in a patient with SLN as assessed with the Rasch-built Overall Disability Scale (RODS).

Secondary objectives: to determine the effect of hydrocortisone treatment on the size of a lipoma in the neck, on the Medical Research Council (MRC) sum score and on specific personalized goals that are important to the patient and the patients' environment (Goal Attainment Scaling (GAS)).

ELIGIBILITY:
The study is especially designed for a specific female patient. The patient is 31 years old at the moment. Since the study is especially designed for this patient, there are no formal inclusion and exclusion criteria. However, the study will be stopped when the patient gets pregnant as this can influence the primary and secondary outcome measures.

Inclusion Criteria:

* N/A

Exclusion Criteria:

* Pregnancy

Min Age: 31 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Rasch-built Overall Disability Scale (RODS) | Baseline to 414 days
  The RODS is a validated 24-items questionnaire to measure the activity and social participation limitations in patients with neuropathy. The questionnaire has a score range of 0 to 100. A higher score means a better outcome (less limitations of the neuropathy)

SECONDARY OUTCOMES:
Size of lipoma | Baseline to 414 days
  The size of the lipoma will be measured with a centimeter by the researcher during hospital visits. The researcher will also take a picture of the lipoma in front of graph paper in a standardized manner. In between hospital visits, the participant will take a picture of the lipoma in front of graph paper.
Medical Research Council (MRC) sumscore | Baseline to 414 days
  The MRC sumscore is a validated tool to measure muscle strength and must be carried out by a physician, nurse, physiotherapist or other professional. The score has a range of 1 to 5. A higher score means a better outcome.
Goal Attainment Scaling (GAS) | Baseline to 414 days
  GAS is an individualized outcome measure in which several personal goals and the corresponding scaling are defined in consultation with the patient. The scaling is standardized, which makes it possible to reliably measure the change in the situation of the patient. The levels range from -3 to +2. A higher level means a better outcome. The predefined personal goals are a measure of the effectivity of the treatment. If possible, three goals will be set.

CONTACTS AND LOCATIONS:
Overall Officials: Laura de Graaff, MD, PhD, Principal Investigator — Department of Internal Medicine - Endocrinology, Erasmus MC, Rotterdam, the Netherlands
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data is available upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available after completion of the study and only upon reasonable request and with permission of the participant.
Access Criteria: A motivated request.